CLINICAL TRIAL: NCT00129688
Title: Comparison of Efficacy, Safety and Economic Outcomes Between Once-Daily Versus Twice-Daily Amikacin in Combination With Cloxacillin in Febrile Neutropenic Children
Brief Title: Once-Daily Amikacin Plus Cloxacillin in Febrile Neutropenic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE44290; 40/2545
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-02

CONDITIONS: Neutropenia; Cancer; Fever
Keywords: febrile neutropenia; once-daily; amikacin; cloxacillin; children
MeSH Terms: conditions — Neutropenia; Neoplasms; Fever; Febrile Neutropenia | interventions — Cloxacillin; Amikacin

INTERVENTIONS:
Drug: cloxacillin and amikacin (once or twice daily dosage)

SUMMARY:
Once-daily dose administration of aminoglycoside in adults is effective and economical. However, its value in febrile neutropenic children, especially in Thailand, is less well researched. In the area where Pseudomonas aeruginosa prevalence in febrile neutropenic children is low, the combination of cloxacillin and amikacin is an appropriate approach. This study would like to compare the efficacy and safety including cost between these two amikacin administrations (once-daily or twice-daily) in combination with cloxacillin as an empirical therapy in febrile neutropenic children.

Hypothesis: Once-daily amikacin plus cloxacillin can be used to treat febrile neutropenic children in Khon Kaen, Thailand.

DETAILED DESCRIPTION:
Fever: a single oral temperature of >/= 38.3 degrees C; or >/= 38.0 degrees C for >/= 1 hour.

Neutropenia: neutrophil count, < 500/cu mm or <1,000/cu mm with a predicted decrease to <500/mm3.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 year - 14 years
* A single oral temperature of >/= 38.3 degrees C; or >/= 38.0 degrees C for >/= 1 hour.
* Neutropenia: neutrophil count, < 500/cu mm or <1,000/cu mm with a predicted decrease to <500/mm3.
* During the course of chemotherapy

Exclusion Criteria:

* History of amikacin or cloxacillin allergy
* Creatinine clearance < 30 ml/min/m2
* Central nervous system infection: meningitis or brain abscess
* History of hearing abnormality
* Severely ill: shock
* Chronic liver diseases or SGPT > 10 times of upper normal limit
* Received aminoglycoside within 14 days prior to enrolment
* Received any intravenous antibiotics within 7 days
* Cancer which is newly diagnosed or relapsed

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166
Dates: Start 2002-04; Study Completion 2004-06

PRIMARY OUTCOMES:
Afebrile within 5 days of the initial treatment regimen
Nephrotoxicity and ototoxicity

SECONDARY OUTCOMES:
Cost difference
Pharmacokinetic parameters of amikacin in these children

CONTACTS AND LOCATIONS:
Overall Officials: Pope - Kosalaraksa, M.D., Principal Investigator — Faculty of Medicine, Khon Kaen University